CLINICAL TRIAL: NCT01614210
Title: Preoperative Window of Endocrine Therapy Provides Information to Increase Compliance
Acronym: POWER PIINC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI57098
Record Dates: First submitted 2012-06-04; First posted 2012-06-07 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Newly Diagnosed Hormone Positive Clinical Stage 1 or 2 Breast Cancer
MeSH Terms: interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All patients enrolled in the study.
  Interventions: Drug: Tamoxifen; Procedure: Breast cancer surgery

INTERVENTIONS:
Drug: Tamoxifen — All patients will take tamoxifen 20 mg po daily for 7 days prior to surgery and for 14 days after surgery.
Procedure: Breast cancer surgery — Breast cancer surgery

SUMMARY:
The purpose of the study is to see if tumors respond to endocrine therapy by taking a total of 21 doses of Tamoxifen before and after surgery. Tamoxifen is currently approved by the FDA (Food and Drug Administration) for use in the treatment of hormone positive breast cancer.

DETAILED DESCRIPTION:
Patients who are eligible (newly diagnosed hormone positive clinical stage 1 or 2 breast cancer) will be approached about the study. If they sign informed consent a prescription for 21 doses of Tamoxifen will be provided. The patient's surgery will be scheduled at a time convenient for the patient and the surgeon. Once the surgery has been scheduled, a medication calendar will be completed that allows the patient to take tamoxifen for 7 days preoperatively with the 7th dose of tamoxifen to coincide with the day before surgery. The patient will continue to take tamoxifen for 2 weeks (14 days) after surgery. Patients will then proceed along normal treatment guidelines. For those needing chemotherapy or radiation therapy, we recommend the long term endocrine therapy start at the conclusion of chemo and/or radiation treatments. For those not going on to any additional therapy, the prescription for endocrine therapy will be written at the initial post-operative visit.

Unstained slides from the formalin-fixed, paraffin-embedded tissue blocks from the patient's breast tissue from which the original diagnosis of breast cancer was made by H&E will be stained for Ki67. After endocrine therapy and subsequent resection, carcinoma will be confirmed by the participating pathologist on H&E, and Ki67 will be performed on unstained slides from a representative tissue block containing invasive carcinoma. The pathologist will circle a designated area of tumor on the H&E slide and both the H&E and immunostained (Ki67) slides will be scanned in a digital imaging device (Aperio XT Scanscope), which quantitatively analyzes the tumor designated by the pathologist with image analysis algorithms. The algorithm accurately detects regions of interest and distinguishes cells and sub-cellular objects within these target regions. It determines morphology and expression profiles per individual cell or cell compartment. For Ki67 analysis, a nuclear Immunohistochemistry (IHC) algorithm will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Diagnosed with hormone receptor positive invasive breast cancer (estrogen receptor (ER) or progesterone receptor (PR) or both >1%) by core needle biopsy
* Clinical American Joint Committee on Cancer (AJCC) 7th edition Stage 1 or 2
* Candidate for surgical therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0,1, or 2
* No chemotherapy or endocrine therapy for breast cancer in last 5 years
* Paraffin fixed core needle tissue block, or biopsy punch available for central analysis for proliferative markers
* Not pregnant or lactating and practicing adequate birth control if premenopausal
* Able and willing to provide informed consent

Exclusion Criteria:

* Prior personal history of uterine cancer
* Prior personal history of stroke or deep vein thrombosis (DVT)
* Current therapy with strong CYP2D6 inhibitors The following medications should not be administered with tamoxifen (21 day treatment period) and will need to be stopped for the designated period of time prior to starting the study tamoxifen.

No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage 0, I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years

Fluoxetine - should be discontinued 30 days prior to starting tamoxifen Paroxetine - should be discontinued 5 days prior to starting tamoxifen Sertraline - should be discontinued 5 days prior to starting tamoxifen Bupropion - should be discontinued 5 days prior to starting tamoxifen

* Concurrent coumarin-type anticoagulation therapy
* Any other contraindications to tamoxifen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Neumayer, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Tamoxifen Pre and Post Breast Surgery: All patients enrolled in the study.
  Tamoxifen: All patients will take tamoxifen 20 mg po daily for 7 days prior to surgery and for 14 days after surgery.
  Breast cancer surgery: Breast cancer surgery
Period: Overall Study
Arm/Group | Tamoxifen Pre and Post Breast Surgery
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tamoxifen Pre and Post Breast Surgery
Number analyzed (Participants) | 52
Age, Continuous [Median (Full Range); unit: years] | 58.5 [38 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Change in Ki67 Expression in Tumors
Description: Demonstrate a significant change in Ki67 expression in tumors with 7 days of pre-surgical tamoxifen.
Time Frame: 7 days
Population: 3 were not evaluable due to rescheduling of surgery; 1 not evaluable due to pharmacy error. 2 patients had no invasive tumor on Ki-67 slides from pretreatment biopsy, and 2 patients had no invasive tumor on post-treatment surgery and were not evaluable.
Measure: Mean (95% Confidence Interval); unit: percentage change in Ki67
Arm/Group | Tamoxifen Pre and Post Breast Surgery
Number analyzed (Participants) | 44
percentage change in Ki67 | -40 [-63 to -29]
Statistical Analysis 1: Comparison: Tamoxifen Pre and Post Breast Surgery; Test type: Other; p = 0.0001, t-test, 1 sided; percentage decrease in Ki67 after 7 days

2. Secondary Outcome: Change in FACT-ES Symptom Scores
Description: Patients were given the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) quality of life assessment at baseline (prior to tamoxifen administration) and again 18 months following breast surgery to assess quality of life. The difference in total score from baseline to 18 months was calculated. The FACT-ES total score ranges from 0-180, with higher scores indicating higher quality of life.
Time Frame: 18 months
Population: Of the 44 patients evaluable for the primary outcome measure, 35 completed both baseline and 18 month FACT-ES assessments
Measure: Mean (95% Confidence Interval); unit: change in units on a scale
Arm/Group | Tamoxifen Pre and Post Breast Surgery
Number analyzed (Participants) | 35
change in units on a scale | -4.53 [-9.68 to 0.62]

3. Secondary Outcome: Number of Participants With Long Term Endocrine Therapy Adherence
Description: For the patient population on this study, endocrine therapy was indicated for 5 years post-surgery according to the current standard of care recommendations for hormone positive breast cancer. Endocrine therapy was prescribed as standard of care as appropriate for each patient's situation. At 18 months post-surgery, patients were evaluated to determine if they were taking their endocrine therapy as prescribed.
Time Frame: 18 months
Population: Of the 52 patients enrolled on the study, 38 patients had data regarding long term endocrine therapy at 18 months post-surgery.
Measure: Number; unit: participants adhering to therapy
Arm/Group | Tamoxifen Pre and Post Breast Surgery
Number analyzed (Participants) | 38
participants adhering to therapy | 33

4. Secondary Outcome: Correlation Between Changes in Ki67 and Symptoms
Description: Evaluate correlation between changes in Ki67 expression and symptom scores. Differences between changes in FACT-ES total score were correlated with changes in Ki67 expression using a the Spearman correlation method and results are expressed as the correlation coefficient.
Time Frame: 7 days
Population: Of the 50 patients enrolled Ki67 measurements were obtained for 44. Of the 44 patients which had a Ki67 result, 43 had both a pre and post symptom score.
Measure: Number; unit: spearman correlation coefficient
Arm/Group | Tamoxifen Pre and Post Breast Surgery
Number analyzed (Participants) | 43
spearman correlation coefficient | -0.02

5. Other Pre Specified Outcome: Change in FACT-ES Symptom Scores
Description: Patients were given the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) quality of life assessment at baseline (prior to tamoxifen administration) and again 7 days following start of tamoxifen to assess quality of life while on tamoxifen. The difference in total score from baseline to 7 days was calculated. The FACT-ES total score ranges from 0-180, with higher scores indicating higher quality of life.
Time Frame: 7 days
Population: Of the 50 patients enrolled, 46 had both pre and post FACT-ES total scores.
Measure: Median (Full Range); unit: change in units on a scale
Arm/Group | Tamoxifen Pre and Post Breast Surgery
Number analyzed (Participants) | 46
change in units on a scale | 1.5 [-54 to 21]

ADVERSE EVENTS:
Arm/Group | Tamoxifen Pre and Post Breast Surgery
Serious Adverse Events (participants affected / at risk) | 1/52
Other Adverse Events (participants affected / at risk) | 42/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamoxifen Pre and Post Breast Surgery (N=52)
Thromboembolic Event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamoxifen Pre and Post Breast Surgery (N=52)
Blurred Vision (Eye disorders) | 3 (3)
Dialated Left Pupil (Eye disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
dry mouth (Gastrointestinal disorders) | 2 (2)
flatulence (Gastrointestinal disorders) | 2 (2)
lip swelling (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (14)
oral pain (Gastrointestinal disorders) | 1 (1)
toothache (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 2 (2)
fatigue (General disorders) | 5 (5)
irritability (General disorders) | 1 (1)
vaginal infection (Infections and infestations) | 1 (1)
bruising (Injury, poisoning and procedural complications) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
akathisia (Nervous system disorders) | 1 (1)
dizziness (Nervous system disorders) | 3 (3)
dysgeusia (Nervous system disorders) | 2 (2)
headache (Nervous system disorders) | 5 (5)
anxiety (Psychiatric disorders) | 1 (1)
insomnia (Psychiatric disorders) | 5 (5)
breast pain (Reproductive system and breast disorders) | 1 (1)
period spotting (Reproductive system and breast disorders) | 1 (1)
vaginal discharge (Reproductive system and breast disorders) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
nasal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1)
flushing (Vascular disorders) | 1 (1)
hot flashes (Vascular disorders) | 19 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes